CLINICAL TRIAL: NCT06341569
Title: Understanding Well-being in Physical Therapy Students: A Multi-Dimensional Analysis of Motivation, Life Satisfaction, and Perceived Academic Quality
Brief Title: Physical Therapy Students: Well-being
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Medicine and Pharmacy "Victor Babes" Timisoara (Other)
Responsible Party: Principal Investigator, Crisan Alexandru Florian, Principal Investigator, University of Medicine and Pharmacy "Victor Babes" Timisoara
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Screening
Other Study IDs: 11/07.03.2024
Record Dates: First submitted 2024-03-14; First posted 2024-04-02 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Anxiety State; Motivation; Life Stress; Sleep, Inadequate
Keywords: Students; Physical Therapy; Anxiety; Motivation; Happiness; Breathing techniques
MeSH Terms: conditions — Anxiety Disorders; Stress, Psychological; Sleep Deprivation

STUDY DESIGN:
Intervention Model Description: This study uses a multiple-group design to investigate various psychosocial aspects of physical therapy students and to explore the potential benefits of breathing techniques as a well-being-promoting intervention. The study involves three groups:
  Intervention group: second-year physical therapy students participating in a 14-week breathing techniques program.
  Control group: second-year physical therapy students who do not participate in the program but complete the same questionnaires.
  Comparison groups: 1st, 2nd, and 3rd year physical therapy students participating in assessments only.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Respiratory breathing techniques group (Experimental): Subjects included in the intervention group will receive a 14 week breathing technique program that will include: different types of breathing techniques (diaphragmatic, pursed-lips, alternate nostril breathing, etc.); progressive muscle relaxation techniques; and medical education about breathing.
  Interventions: Other: Respiratory breathing techniques group
- Control group (No Intervention): Second-year physical therapy students that do not want to participate in the breathing technique program and will complete only the questionnaires.

INTERVENTIONS:
Other: Respiratory breathing techniques group — Target group: subjects in the respiratory breathing techniques group. Program duration: the program lasts for 14 weeks.
  Breathing techniques: the program includes various breathing exercises, including:
  Diaphragmatic breathing teaches participants to breathe deeply, engaging the diaphragm muscle, which can improve lung capacity and relaxation.
  Pursed-lips breathing: this technique involves inhaling through the nose and exhaling slowly through pursed lips, which can help slow down breathing and manage shortness of breath.
  Alternate nostril breathing: this technique involves closing one nostril while inhaling and exhaling through the other nostril alternately.
  Relaxation techniques: the program incorporates progressive muscle relaxation techniques. This involves progressively tensing and relaxing different muscle groups.
  Medical education: topics like the anatomy of the respiratory system, the importance of proper breathing, potential benefits of specific breathing exercises.
  Arms: Respiratory breathing techniques group

SUMMARY:
This study aims to explore various psychosocial aspects and the potential benefits of respiratory techniques for physical therapy students.

DETAILED DESCRIPTION:
Understanding the psychosocial state of academic students has become a primary concern in contemporary educational research and practice. As students go through the challenges of higher education, factors such as motivation, life satisfaction, and happiness play crucial roles in shaping their academic experiences and outcomes. Therefore, researchers have increasingly turned their attention to studying these elements in order to gain insight into the overall state of students and inform strategies designed to create positive educational outcomes.

The implications of studying motivation, life satisfaction, and happiness among academic students are far-reaching. By gaining a deeper understanding of these psychosocial elements, educators and policymakers can develop interventions and programs designed to cultivate positive learning environments that support students' psychological well-being and academic success. For example, strategies that enhance intrinsic motivation, such as promoting autonomy and providing meaningful learning opportunities, can lead to improved engagement and academic achievement. Similarly, initiatives that promote a sense of belonging and social support can improve students' overall life satisfaction and happiness.

Thus, this study aims to explore various psychosocial aspects and the potential benefits of respiratory techniques for physical therapy students.

ELIGIBILITY:
Inclusion Criteria:

Students: enrolled in the physical therapy study program (year I, II and III) Age: > 18 years Ability to understand and follow instructions Availability to provide informed consent.

Exclusion Criteria:

Pre-existing medical conditions: uncontrolled medical conditions (cardiovascular disease, severe respiratory problems) Use of psychotropic drugs: drugs that could significantly affect mood, anxiety level, or sleep quality.

Pregnancy: due to potential physiological changes that could influence the results of the study.

Inability to comply with study requirements: these could include completing questionnaires and participating in the respiratory techniques program (if part of the intervention group).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2024-05-09 (Actual); Primary Completion 2024-08-29 (Actual); Study Completion 2024-10-30 (Actual)

PRIMARY OUTCOMES:
Assessing intrinsic and extrinsic motivation levels among physical therapy students. | At the beginning of the study
  The Motivational Styles Questionnaire (MSLQ) assesses students' intrinsic and extrinsic motivation levels. The MSLQ does not have a standard range of minimum and maximum values. Higher scores on intrinsic motivation indicate a better outcome, reflecting a higher level of internal motivation. Conversely, higher scores on extrinsic motivation may suggest a reliance on external rewards or pressures, which could indicate a less favorable outcome.
Assessing the happiness levels of the students participating in the study. | At the beginning of the study
  The Oxford Happiness Questionnaire evaluates happiness levels. It ranges from 1 to 6. Higher scores on the Oxford Happiness Questionnaire indicate a better outcome, reflecting higher happiness and life satisfaction levels.
Assessing the positive and negative emotional states of the students participating in the study. | At the beginning of the study
  The PANAS-GEN Questionnaire measures positive and negative expressions to provide insights into emotional states. It ranges from 1 to 5. Higher scores on positive expressions indicate a better outcome, reflecting higher positive emotions. Conversely, higher scores on negative expressions may suggest a less favorable outcome, indicating higher levels of negative emotions.
Assessing the well-being of the students participating in the study. | At the beginning of the study
  The RYFF Psychological Well-being Questionnaire assesses different aspects of psychological well-being among students. The RYFF Psychological Well-being Questionnaire typically ranges from 1 to 6. Higher scores on the RYFF Psychological Well-being Questionnaire indicate a better outcome, reflecting higher levels of psychological well-being.
Assessing the overall life satisfaction levels of the students participating in the study. | At the beginning of the study
  The Satisfaction with Life Questionnaire evaluates overall life satisfaction. It ranges from 1 to 7. Higher scores on the Satisfaction with Life Questionnaire indicate a better outcome and reflect higher levels of life satisfaction.
Assessing the subjective happiness levels of the students participating in the study. | At the beginning of the study
  The Subjective Happiness Scale assesses subjective happiness levels. It ranges from 1 to 7. Higher scores on the Subjective Happiness Scale indicate a better outcome, reflecting higher levels of subjective happiness.
Assessing the sleep quality of the students participating in the study. | At the beginning of the study
  The Pittsburgh Quality of Sleep Index (PSQI) evaluates the sleep quality of the participants. It ranges from 0 to 21. Lower scores on the PSQI indicate a better outcome, reflecting higher sleep quality.
Assessing the worry and anxiety levels of the students participating in the study. | At the beginning of the study
  The Penn State Worry Questionnaire (PSWQ) assesses students' worry and anxiety levels. It ranges from 1 to 5. Lower scores on the PSWQ indicate a better outcome, reflecting lower levels of worry and anxiety.
Assessing the effects of the respiratory techniques program on the intrinsic and extrinsic motivation levels of the students participating in the study. | 14 weeks after the beginning of the study
  Comparison of the MSLQ baseline scores before and after 14 weeks of the respiratory techniques program. Higher scores on intrinsic motivation indicate a better outcome, reflecting a higher level of internal motivation. Conversely, higher scores on extrinsic motivation may suggest a reliance on external rewards or pressures, which could indicate a less favorable outcome.
Assessing the effects of the respiratory techniques program on the happiness levels of the students participating in the study. | 14 weeks after the beginning of the study
  Comparison of the Oxford Happiness Questionnaire baseline scores before and after 14 weeks of the respiratory techniques program. Higher scores on the Oxford Happiness Questionnaire indicate a better outcome, reflecting higher happiness and life satisfaction levels.
Assessing the effects of the respiratory techniques program on the students' positive and negative emotional states. | 14 weeks after the beginning of the study
  Comparison of the PANAS-GEN Questionnaire baseline scores before and after 14 weeks of the respiratory techniques program. Higher scores on positive expressions indicate a better outcome, reflecting higher positive emotions. Conversely, higher scores on negative expressions may suggest a less favorable outcome, indicating higher levels of negative emotions.
Assessing the effects of the respiratory techniques program on the students' well-being. | 14 weeks after the beginning of the study
  Comparison of the RYFF Psychological Well-being Questionnaire baseline scores before and after 14 weeks of the respiratory techniques program. Higher scores on the RYFF Psychological Well-being Questionnaire indicate a better outcome, reflecting higher levels of psychological well-being.
Assessing the effects of the respiratory techniques program on the overall life satisfaction levels of the students participating in the study. | 14 weeks after the beginning of the study
  Comparison of the Satisfaction with Life Questionnaire baseline scores before and after 14 weeks of the respiratory techniques program. Higher scores on the Satisfaction with Life Questionnaire indicate a better outcome, reflecting higher levels of life satisfaction.
Assessing the effects of the respiratory techniques program on the subjective happiness levels of the students participating in the study. | 14 weeks after the beginning of the study
  Comparison of the Subjective Happiness Scale baseline scores before and after 14 weeks of the respiratory techniques program. Higher scores on the Subjective Happiness Scale indicate a better outcome, reflecting higher levels of subjective happiness.
Assessing the effects of the respiratory techniques program on the quality of sleep of the students participating in the study. | 14 weeks after the beginning of the study
  Comparison of the Pittsburgh Quality of Sleep Index (PSQI) baseline scores before and after 14 weeks of the respiratory techniques program. Lower scores on the PSQI indicate a better outcome, reflecting higher sleep quality.
Assessing the effects of the respiratory techniques program on the worry and anxiety levels of the students participating in the study. | 14 weeks after the beginning of the study
  Comparison of the Penn State Worry Questionnaire (PSWQ) baseline scores before and after 14 weeks of the respiratory techniques program. Lower scores on the PSWQ indicate a better outcome, reflecting lower levels of worry and anxiety
Adherence to breathing exercises at 12-month follow-up | 12 months after the end of the intervention
  Adherence will be assessed using a structured self-report questionnaire developed for this study. Key variables include: weekly frequency, session duration, technique used, barriers, and perceived utility. A composite dose index (frequency × duration) and binary adherence variable will be calculated. Full questionnaire, codebook, and scoring instructions are available at: https://doi.org/10.17605/OSF.IO/T9XAP
Coping strategies assessed with the COPE at 12-month follow-up | 12 months after the end of the intervention
  Coping will be measured using the COPE inventory (50-item version). The scale includes multiple subscales such as active coping, emotional support, denial, acceptance, planning, and others. Subscale scores will be computed according to the scoring manual.
Self-esteem assessed with the Rosenberg Self-Esteem Scale at 12-month follow-up | 12 months after the end of the intervention
  Self-esteem will be measured using the Rosenberg Self-Esteem Scale (RSES), a 10-item validated questionnaire. Higher total scores indicate higher self-esteem.
Perceived psychological benefit of breathing practice at 12-month follow-up | 12 months after the end of the intervention
  Psychological benefit will be evaluated using four Likert-scale items measuring perceived improvement in stress, sleep, positivity, and worry. A composite mean score will be calculated (Perceived_benefit_mean). Instrument details and scoring instructions are available at: https://doi.org/10.17605/OSF.IO/T9XAP

CONTACTS AND LOCATIONS:
Overall Officials: Alexandru Florian Crisan, PhD, Principal Investigator — University of Medicine and Pharmacy "Victor Babes" Timisoara
Locations (1):
- University of Medicine and Pharmacy Victor Babes Timisoara, Timișoara, Timiș County, Romania

REFERENCES:
- [Derived] Crisan AF, Pescaru CC, Maritescu A, Carunta V, Stoicescu ER, Oancea C, Amaricai E, Onofrei RR. A 14-week structured breathing program: an investigation into its impact on psychological health parameters in university students. BMC Public Health. 2025 Apr 14;25(1):1395. doi: 10.1186/s12889-025-22585-8. PMID 40229773